CLINICAL TRIAL: NCT07072052
Title: Oxford Luteal Dysfunction and Placental Insufficiency Study
Acronym: OxLuPIn
Status: Not yet recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: PID17872
Record Dates: First submitted 2025-06-25; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Pre-eclampsia
Keywords: corpus luteum; pre-eclampsia; early pregnancy; prognostic marker; risk stratification
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All consenting participants will undergo venepuncture on two occasions: at <8 weeks' gestation (research visit 1) and at 10-14 weeks' gestation (research visit Blood will be taken in the following formats and retained: EDTA plasma, Silica serum, SST serum, Lithium heparin, Citrate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy pregnant volunteers: Healthy pregnant volunteers at <8 completed weeks of gestation (i.e., up to 7 weeks and 6 days' gestation)
  Interventions: Other: No intervention planned

INTERVENTIONS:
Other: No intervention planned — No interventions planned

SUMMARY:
High blood pressure (BP) affects approximately 1 in 10 pregnancies. About half of women with high blood pressure in pregnancy develop a serious complication called preeclampsia, which kills over 70,000 women and 500,000 babies every year worldwide. Despite its devastating impact, scientists know little about preeclampsia prevention or treatment. Research has shown that preeclampsia results mainly from an abnormal attachment of the placenta to the lining of the womb. In the first 8 weeks of pregnancy, placental attachment depends on the release of hormones (for example, progesterone) by a gland in the ovary called the corpus luteum. Low blood levels of progesterone in early pregnancy are associated with a reduced chance of having a live baby and higher risk of miscarriage. Giving progesterone to women at risk of miscarriage in early pregnancy reduces their chance of developing preeclampsia by nearly 40%. These results highlight the crucial role of the corpus luteum in normal pregnancy, but there is a need for high-quality studies to identify women whose corpus luteum may be defective. Giving these women medicines to treat corpus luteal defects may lead to normal attachment of the placenta, reducing the risk of pregnancy complications such as preeclampsia. The investigators propose a study that will investigate whether ultrasound features of the corpus luteum and blood and urine levels of corpus luteal hormones may predict preeclampsia.

DETAILED DESCRIPTION:
The corpus luteum (CL), formed in the ovary after ovulation, secretes a range of molecules (e.g., oestradiol, progesterone, vascular endothelial growth factor [VEGF], relaxin-2) that regulate embryo implantation and placentation.1 Without a CL, early pregnancy invariably fails, unless women receive exogenous hormone replacement.2 After 8 weeks of pregnancy, the placenta takes over endogenous hormone synthesis from the CL, ensuring pregnancy maintenance until birth; this is termed the luteo-placental shift.2 3 Placental maladaptation is the principal driver of preeclampsia, a pregnancy complication that kills >70,000 women and 500,000 babies annually worldwide.4 Despite its catastrophic effects, there remains a paucity of interventions to prevent or treat preeclampsia. The best tool currently available to predict preeclampsia in the index pregnancy is a validated algorithm which can only be used at 10-14 weeks (the Fetal Medicine Foundation [FMF] Preeclampsia prediction tool, whose positive predictive value is 90%).5

The role of the CL in orchestrating placentation has recently gained prominence following a huge rise in frozen embryo transfer (FET) treatment in assisted conception.6 There are different methods of preparing the endometrium for FET. These include unmedicated regimens, relying on the woman's menstrual cycle to time embryo transfer; and medicated protocols, involving the administration of oestradiol and progesterone before embryo transfer.7 The latter suppresses the pituitary gland, preventing ovulation and the formation of a CL. Uniquely, pregnancies resulting from medicated FET cycles are the only gestations capable of reaching viability without a CL, and are only able to progress because of early hormone replacement.8

Pregnancies without a functioning CL exhibit more than double the odds of preeclampsia (odds ratio [OR] 2.13, 95% confidence interval [CI] 1.89-2.38; 4 studies; n = 22,856 women) versus pregnancies with a functioning CL,8 highlighting a crucial role of the CL in preventing placental maladaptation. Our previous work has elucidated this role by showing a strong association between low luteal serum progesterone and reduced odds of live birth (adjusted OR 0.41, 95% CI 0.18-0.91).9 10 We have also demonstrated that administering exogenous progesterone in early pregnancy significantly reduces the incidence of preeclampsia (risk ratio [RR] 0.61, 95% CI 0.41-0.92; 3 randomised controlled trials [RCTs]; I2 = 0%; n = 5,267 women).11 These findings provide a strong signal that luteal phase insufficiency plays a fundamental role in placental maladaptation, yet crucially it appears amenable to exogenous rescue.

Case-control evidence suggests an association between low serum levels of corpus luteal products, including progesterone and relaxin-2, and the risk of preeclampsia, although data remain scarce and of low quality.12 13 In addition, current practice involves screening women in early pregnancy for their risk of preeclampsia based on their history, yielding a detection rate that is at most 30%.14 Identifying blood and ultrasound markers in early pregnancy associated with the risk of developing preeclampsia later on would allow to develop diagnostic tests and therapeutic targets to prevent preeclampsia.

Therefore, this study aims to establish the association between early serum and ultrasound markers of corpus luteal function and pregnant women's risk of developing preeclampsia. By focusing on recruiting women in very early gestation (<8 weeks), we aim to develop a set of prognostic markers which will help to better identify women at high risk of developing preeclampsia as early as possible. This will allow for better risk stratification in this population, and for future trials investigating interventions to prevent preeclampsia from early gestation rather than at 12 weeks (e.g., when aspirin is currently commenced) which may be too late to effectively correct placental maladaptation.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give written informed consent for participation in the study.
* Female, aged 16 years or above. As in vitro fertilisation is not undertaken in women younger than 18 years, those with pregnancies resulting from natural cycle frozen embryo transfer will be aged 18 years or above.
* Pregnancy <8 completed weeks of gestation (i.e., up to 7 weeks and 6 days' gestation).
* Conception through any of the following means: unassisted ("natural"), ovulation induction (with clomifene citrate, letrozole or gonadotropin injections, including trigger injection), intrauterine insemination (with or without ovulation induction, including trigger injection), or natural cycle frozen embryo transfer.
* Intrauterine viable pregnancy confirmed on research ultrasound scan.
* Intention to deliver at Oxford University Hospitals.

Exclusion Criteria:

* Unable to read, or to understand written or spoken English.
* Vaginal bleeding at first visit.
* Miscarriage at first visit, defined as fetal crown-rump length of 7 mm or longer with no visible heartbeat, OR gestational sac with a mean of 25 mm or greater in diameter with no visible fetal pole on ultrasonography.
* Evidence of ectopic pregnancy at first visit.
* Multiple pregnancy.
* Uterine pathology (e.g., uterine polyp, fibroid, septate uterus, uterus didelphys, bicornuate uterus, unicornuate uterus).
* Fresh in vitro fertilisation.
* Donor oocyte in vitro fertilisation.
* Frozen embryo transfer using hormone replacement therapy for endometrial preparation.
* Participation in any concurrent trials of medicinal products in pregnancy.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy pregnant volunteers at <8 completed weeks of gestation (i.e., up to 7 weeks and 6 days' gestation)
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between early luteal secretory product levels and preeclampsia risk | Collected data and samples will be analysed blindly throughout the study and compared between the two main time points: <8 weeks' gestation (research visit 1) 10-14 weeks' gestation (research visit 2)
  To evaluate the correlation between individual levels of corpus luteum secretory products at <8 weeks' gestation: progesterone (ng/mL), oestradiol (pmol/mL), vascular endothelial growth factor (VEGF) and Relaxin-2, measured in serum/plasma and the predicted probability (%) of developing preeclampsia at 10-14 weeks' gestation using the validated Fetal Medicine Foundation Preeclampsia Prediction Algorithm.
Correlation between luteal ultrasound features and preeclampsia risk | Collected data and samples will be analysed throughout the study and compared between the two main time points: <8 weeks' gestation (research visit 1) 10-14 weeks' gestation (research visit 2)
  Evaluate the correlation between ultrasound imaging characteristics (corpus luteum size and vascularity index measured by power Doppler), and the calculated probability (%) of developing preeclampsia, as predicted by the Fetal Medicine Foundation Preeclampsia Prediction Algorithm at 10-14 weeks' gestation.

SECONDARY OUTCOMES:
Correlation between corpus luteal function and placental volume at 10-14 weeks | Visit 1 (<8 weeks) and Visit 2 (10-14 weeks)
  To determine the correlation between corpus luteum function (progesterone (ng/mL), oestradiol (pmol/mL), vascular endothelial growth factor (VEGF) and Relaxin-2, measured in serum/plasma and ultrasound imaging characteristics of corpus luteum size and vascularity) and placental volume (cm³) measured by 3D ultrasound at 10-14 weeks' gestation.
Correlation between corpus luteum function and placental vascularity index at 10-14 weeks | Visit 1 (<8 weeks) and Visit 2 (10-14 weeks)
  To determine the correlation between corpus luteum function <8 weeks (progesterone (ng/mL), oestradiol (pmol/mL), vascular endothelial growth factor (VEGF) and Relaxin-2, measured in serum/plasma and ultrasound imaging characteristics of corpus luteum size and vascularity) and placental vascularity index (from power Doppler ultrasound) at 10-14 weeks' gestation.
Incidence of pre-eclampsia | These outcomes will be collected via telephone calls and medical records at the following weeks of pregnancy: Weeks 18-21 (usual care [UC] visit 1 - routine hospital attendance for anomaly scan), delivery and up to 4-6 weeks post delivery
  Proportion (%) of participants who develop preeclampsia.
Incidence of fetal growth restriction | These outcomes will be collected via telephone calls and medical records at the following weeks of pregnancy: Weeks 18-21 (usual care [UC] visit 1 - routine hospital attendance for anomaly scan), delivery and up to 4-6 weeks post delivery
  Proportion (%) of pregnancies affected by fetal growth restriction (FGR), defined as estimated fetal weight <10th percentile or abdominal circumference <3rd centile, or <10th centile with Doppler abnormalities
Incidence of preterm birth | At delivery (≥24 weeks)
  Proportion (%) of live births occurring before 37+0 weeks' gestation.
Birth weight | At delivery
  Mean birth weight in grams among live births.
Association between corpus luteal function and placental dysfunction | These outcomes will be collected via telephone calls and medical records at the following weeks of pregnancy: Weeks 18-21 (usual care [UC] visit 1 - routine hospital attendance for anomaly scan), delivery and up to 4-6 weeks post delivery
  This outcome represents a composite of clinically relevant adverse pregnancy outcomes associated with impaired placentation related to corpus luteum function (progesterone (ng/mL), oestradiol (pmol/mL), vascular endothelial growth factor (VEGF) and Relaxin-2, measured in serum/plasma and ultrasound imaging characteristics of corpus luteum size and vascularity) The composite includes any of the following conditions: gestational hypertension, preeclampsia, fetal growth restriction, and preterm birth. % of participants experiencing any of the above conditions

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Melo, MD PhD MRCOG, Principal Investigator — Nuffield Department of Women's and Reproductive Health
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided